CLINICAL TRIAL: NCT02064660
Title: An Integrative Medical Approach of Acupoint Stimulation for Children With Myopia : A Pilot Study
Brief Title: The Efficacy and Safety of Periocular Acupoint Stimulation on Myopia Progression in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Principal Investigator, Ki-Bong, Kim, Assistant Professor, Korean Medicine Hospital of Pusan National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: blueicek
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Myopia
Keywords: Myopia; Children; Acupressure; Refractive error; Axial length; Korean medicine
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): A series of acupressure sessions within six months from the baseline
  Interventions: Device: massager

INTERVENTIONS:
Device: massager — The patients will be doing self-stimulation using acupressure device, The acupuncture treatment will be applied two times per day for six months. Acupressure divice will stimulate for 14 minutes. Examples of acupuncture points to be used might include GB1, GB14, TE23, ST1, ST2, BL01, BL02, the Extra-point Tae-yang, In-dang.
  Other Names: proprietary name : Nurieye-1

SUMMARY:
Myopia is widely one of the three commonly detected refractive errors. Myopia is usually managed by correction through glasses or contact lenses. Other alternative available include surgery, drugs and acupuncture. There are various therapeutic approaches and different points can be used in acupuncture treatment for myopia, such as auricular acupuncture, acupressure body acupuncture. However, the mechanism of acupuncture therapy for myopia is largely unknown. Furthermore, little information exists regarding the effects and safety of acupuncture for degenerative myopia in children.

The investigators aimed to assess the overall effectiveness, safety of periocular acupressure for children with myopia

The hypotheses of this study are as follows:

Periocular acupressure is effective for myopia progression delay.

The study aims to include 56 participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-12 years
* Spherical equivalent greater than -5D
* Individuals without strabismus, anistopia
* Willingness to participate in the study

Exclusion Criteria:

* The presence of a related disease such as cataract, glaucoma, or other eye disease.
* Individuals who were received ocular or scalp trauma.
* Individuals who were received ocular surgery and had ocular wound.
* Individuals who were adapted bifocal lense.
* Individuals suffering fever or bad conditions.
* Individuals suffering systemic or neurologic disease.
* Indibiduals who were receiving other therapy during the period of study
* Individuals who did not comply with the treatment which affected myopia progression.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Refractive error | 6 months
  Change from baseline in the refractive erros will be used.

SECONDARY OUTCOMES:
Axial length | 6 months
  Change from baseline in the axial length will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Ki-bong Kim, Principal Investigator — Pusan National University Korean Medicine Hospital
Locations (1):
- Pusan National University Korean Medicine Hospital, Yangsan, Gyeongsangnam-do, South Korea